CLINICAL TRIAL: NCT04084236
Title: The Effects of Transcutaneous Electrical Nerve Stimulation on People With Knee Osteoarthritis (OA) and or Chronic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Omron Healthcare Co., Ltd. (Industry)
Collaborators: Western Michigan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HDV-CDD-180139
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Knee Pain
MeSH Terms: interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active TENS (Active Comparator)
  Interventions: Device: electrical stimulation
- Sham TENS (Sham Comparator)
  Interventions: Device: Sham

INTERVENTIONS:
Device: electrical stimulation — electrical stimulation
  Arms: Active TENS
Device: Sham — no stimulation
  Arms: Sham TENS

SUMMARY:
The purpose of this study is to evaluate the effect of TENS at the knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female between the ages of 45 years or older
* Ultrasonography scale of 0-3 for grading of primary Knee OA of the knee(s)
* Pain perceived as a minimum of 3/10 on a 0-10 pain scale with 24 hours of the each visit
* No phobia of electrical stimulation
* No pain or anti-inflammatory medication will be taken during study
* OA and or Chronic knee pain, Injury/pain that began minimum of 6- weeks before the beginning of the study.

Exclusion Criteria:

* Pregnancy
* Diabetes Mellitus
* Neuropathy
* Smoker
* Uncontrolled HTN
* Past surgery in the region to be treated by TENS or had received an intra-articular corticosteroid or hyaluronic acid injection within 6 months prior to enrollment
* Arthritis (RA) in the area to be treated by TENS
* Allergic to tape/electrodes
* Dementia
* History of knee joint replacement or tibial osteotomy
* Undergoing physical therapy
* Any major joint pain (e.g., back, hip, or ankle) that could limit functional ability
* Contraindications to TENS (pacemakers, dermatological conditions, and abnormal sensation in the knees)
* Severe medical or neurological conditions (e.g. Chronic obstructive pulmonary disease, cardiovascular disease, arteriosclerosis obliterans, cerebrovascular accident, lumber disc, herniation, and rheumatoid arthritis)
* The subject does not utilize stairs in daily living
* The subject is unable to walk without ambulatory assistive devices.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
stair climb test | 2 hours
  An 11-step stairway with a step height of 17 cm will be used. Participants will begin with both feet on the bottom landing, then ascend and descend the stairway as fast as possible, and finally stop with both feet back on the bottom landing while using a handrail support, if required. Time recording will be started when the participant is signalled to start and ended when the participant returns with both feet on the ground.
timed Up and Go test (TUG) | 2 hours
  The participant will sit down at first and then stand up when given the signal to start. As fast as possible, the participant will walk 3 meters toward a cone on the floor, circle it, walk back 3 more meters toward a chair, and finally sat down. Timing begins on the signal to start and ends when the participant completely sits down with their back resting on the backrest of the chair.
6-minute walk test (6MWT) | 2 hours
  In the 6MWT, the participants will walk as far as they could within 6 minutes. They will not be allowed to carry a watch or provided feedback during the trial. Although rest periods are allowed, time recording will continue. The participants will be provided encouragement at 1-minute intervals.
VAS(Visual Analog Scale score) for knee pain | 2 hours
  The mean knee pain during the stair climb test, TUG test, and 6MWT will be measured using the VAS. Participants will record their level of knee pain by drawing a vertical mark between the ends of a 10-cm horizontal line. The 0-cm end and the 10-cm end represented no pain and the most extreme pain, respectively.
The Knee injury and Osteoarthritis Outcome Score (KOOS) | 2 hours
  The Knee injury and Osteoarthritis Outcome Score (KOOS) was developed as an extension of the WOMAC Osteoarthritis Index with the purpose of evaluating short-term and long-term symptoms and function in subjects with knee injury and osteoarthritis. The KOOS holds five separately scored subscales: Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL).
Perceived Competence Scale (PCS) questionnaire | 2 hours
  The Perceived Competence Scale (PCS) concerns feelings about behaving in healthy ways. This is a short 4-item questionnaire that assesses the degree to which participants feel confident about being able to make (or maintain) a change toward a healthy behavior, participate in a health-care program, or carry out a treatment regimen/physical tests.
The Hospital Anxiety and Depression Scale (HADS) | 2 hours
  HADS was found to perform well in assessing the symptom severity of anxiety disorders and depression in in the general population. The sensitivity and specificity for both HADS-A and HADS-D of approximately 0.80. The questionnaire comprises seven questions for anxiety and seven questions for depression.

SECONDARY OUTCOMES:
2-step test | 2 hours
  Gait stride length is measured to assess walking ability, including muscle strength, balance, and flexibility of the lower limbs. The starting line is determined, and participants stand with the toes of both feet behind this line. They take 2 long steps (as long as possible) and then align both their feet. Subsequently, the length of the 2 steps from the starting line to the toes is measured.
stand-up test | 2 hours
  The participant will stand up on 1 or both legs from a seat at a specified height. For this test, 4 seats are set up at different heights (40, 30, 20, and 10 cm). First, the participants will sit on the 40-cm high seat with arms folded. If they can stand up on both legs, they then attempt to stand on 1 leg. If they can stand up on both their right and left legs, they pass the height level. The participants then repeat the trial at the next seat height, and the trials will be performed in the order of descending height.
Knee extensor strength | 2 hours
  The maximum isometric knee extensor strengths will be measured using a handheld dynamometer (HHD), which is the validated method in a previous research on elderly individuals who are prone to falls.17 The maximum force will be recorded in Newtons (N), and testing will be repeated for 2 measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Omron healthcare Co.,Ltd., Mukō, Japan